CLINICAL TRIAL: NCT00896129
Title: Mid-to Long-Term Outcomes in Chronic Myeloid Leukemia Patients With Complete Cytogenetic Response Treated With Imatinib as First Line Therapy: Health-Related Quality of Life, Symptom Burden and Adherence to Therapy Issues.
Brief Title: Mid-to Long-Term Outcomes in Chronic Myeloid Leukemia (CML) Patients With Complete Cytogenetic Response After Imatinib as First Line Therapy
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: QOL-CML0208
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Health Outcomes Research; CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population
  Interventions: Other: HRQOL Survey Packet

INTERVENTIONS:
Other: HRQOL Survey Packet — Questionnaires

SUMMARY:
Rationale: At present, virtually no evidence exists regarding mid to long-term patient-reported health outcomes (e.g., health related quality of life-HRQOL) of CML patients treated with Imatinib.

Purpose: the results of this research will provide preliminary evidence-based data on an number of issues from the patients' perspective, including adherence to therapy issues.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary: to investigate a number of mid to long-term HRQOL issues in Chronic Myeloid Leukemia (CML) patients with complete cytogenetic response treated with Imatinib as First Line Therapy.

Secondary evaluation of:

* Psychological wellbeing.
* Fatigue.
* Adherence to therapy issues.
* Symptom burden.
* Possible association between social-demographic and clinical variables with patient reported health outcomes.

OUTLINE:This is a multicenter study.

SAMPLE SIZE:

Sample size estimation has not been performed considering the nature of the study and the lack of preliminary data to hypothesize the number of possible eligible patients in each center.

DURATION OF THE STUDY:

The recruitment period is estimated in approximately 6 to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years.
* CML patients meeting the following criteria:

  * Started IM therapy in the early chronic phase (ECP).
  * Have been undergoing treatment with IM, as first line therapy, for at least three years regardless of the current prescribed dose of IM.
  * In complete cytogenetic response (CCgR) and no clinical evidence of disease progression to accelerated phase (AP) or blast crisis (BC).
* Able to read and write Italian.
* Freedom from psychiatric conditions that may confound HRQOL evaluation.
* Informed consent provided.

Exclusion Criteria:

* CML patients who were initially diagnosed in the AP or BC or those who started therapy with IM in the late chronic phase (LCP).
* Having received any kind of treatment prior to IM therapy (except for hydroxyurea and/or anagrelide).
* Patients with a new primary malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult CML patiens under Imatinib treatment for at least three years
Sampling Method: Non-Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number of mid to long-term HRQOL issues in Chronic Myeloid Leukemia (CML) patients with complete cytogenetic response treated with Imatinib as First Line Therapy. | By the end of the study.

SECONDARY OUTCOMES:
Psychological wellbeing. | By the end of the study.
Fatigue. | By the end of the study.
Adherence to therapy issues. | By the end of the study.
Symptom burden. | By the end of the study.
Possible association between socio-demographic and clinical variables with patient reported health outcomes. | By the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Efficace, PhD, Study Chair — GIMEMA Foundation
Locations (25):
- Italy (25):
  - Ist.Ematologia e Oncologia Medica L.e A. Seragnoli, Bologna, Bologna
  - Serv. di Ematologia Ist. di Ematologia ed Endocrinologia, Sassari, Sassari
  - Nuovo ospedale "Torrette", Ancona
  - Unità Operativa Ematologica - Università degli Studi di Bari, Bari
  - Ospedali Riuniti, Bergamo
  - Sezione di Ematologia e Trapianti Spedali Civili, Brescia
  - Azienda ASL di Cagliari, Cagliari
  - Ospedale Ferrarotto, Catania
  - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro
  - Sez.Ematologia e Dip. scienze Biomediche Arcispedale S. Anna, Ferrara
  - Clinica Ematologica - Università degli Studi, Genova
  - Ematologia 1 - Centro Trapianto di Midollo, Milan
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II", Napoli
  - Ospedale S. Luigi Gonzaga, Orbassano
  - Ospedale Cervello, Palermo
  - Azienda ASL di Pescara, Pescara
  - Università di Pisa, Azienda Ospedaliera Pisana, Pisa
  - Ospedale S.Maria delle Croci, Ravenna
  - Ospedali Riuniti - Div. di Ematologia, Reggio Calabria
  - Università La Sapienza, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - U.O. Ematologia, Azienda Ospedaliera Universitaria Senese, Siena
  - Azienda USL 9 Treviso - U.O. di Ematologia, Treviso
  - Policlinico G.B. Rossi, Verona

REFERENCES:
- [Background] Efficace F, Baccarani M, Breccia M, Alimena G, Rosti G, Cottone F, Deliliers GL, Barate C, Rossi AR, Fioritoni G, Luciano L, Turri D, Martino B, Di Raimondo F, Dabusti M, Bergamaschi M, Leoni P, Simula MP, Levato L, Ulisciani S, Veneri D, Sica S, Rambaldi A, Vignetti M, Mandelli F; GIMEMA. Health-related quality of life in chronic myeloid leukemia patients receiving long-term therapy with imatinib compared with the general population. Blood. 2011 Oct 27;118(17):4554-60. doi: 10.1182/blood-2011-04-347575. Epub 2011 Jul 12. PMID 21750313
- See also: Related Info — http://www.gimema.it